CLINICAL TRIAL: NCT04513860
Title: Cenobamate Expanded Access Program (EAP)
Status: Approved for marketing | Type: Expanded Access
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C013, C017, C021 EAP
Record Dates: First submitted 2020-08-04; First posted 2020-08-14 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Partial Epilepsy
Keywords: Partial onset seizures; Treatment resistant; Partial epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Cenobamate

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: YKP3089 — Capsule, dose to be titrated Tablet, dose to be titrated
  Other Names: Cenobamate

SUMMARY:
This Cenobamate Expanded Access Program (EAP) is designed to continue providing treatment with Cenobamate (YKP3089) to patients with partial-onset epilepsy that were enrolled in the SK Life Science clinical trial YKP3089C013, YKP3089C017 or YKP3089C021.

DETAILED DESCRIPTION:
This Expanded Access Program (EAP) is designed to provide access to an unlicensed drug that is approved in the United States for the treatment of a serious or life-threatening condition. This EAP will be sponsored by SK Life Science Inc. and managed by WEP Clinical. Cenobamate is approved for the treatment of partial onset seizures in adults in United States. The attached US Label (appendix 1) provides the most recent guidance for use of cenobamate.

The objective of this EAP is to continue providing treatment with Cenobamate (YKP3089) to patients with partial-onset epilepsy that were enrolled in the SK Life Science clinical trial YKP3089C013, YKP3089C017 or YKP3089C021. Access to Cenobamate under this guideline is considered a treatment scenario and is not a clinical trial.

Epilepsy is a symptom of a neurological problem that causes sudden, brief seizures. It leads to an increased risk of injury from accidents, an increased rate of mortality, and has a significant impact on quality of life. Epilepsy can occur as a result of a neurological injury, a structural brain lesion, as a part of many systemic medical diseases or may be generic in origin. The incidence of having epilepsy during a lifetime is between 2-5%. Available medications control seizures in 50% of patients and decrease seizure incidence in 75%. The remainder continued to have unacceptable number of seizures, side effects, and psychiatric symptoms. The high treatment failure may be the result of inadequate efficacy or intolerable side effects that lead to poor compliance.

Cenobamate is a novel small molecule that is an antiepileptic agent for partial onset seizures. The precise mechanism by which cenobamate exerts its therapeutic effects in patients with partial-onset seizures is unknown. Cenobamate has been demonstrated to reduce repetitive neuronal firing by inhibiting voltage-gated sodium currents. It is also a positive allosteric modulator of the γ-aminobutyric acid (GABAA) ion channel.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients currently enrolled in one of the following SK life science studies: YKP3089C013, YKP3089C017 or YKP3089C021.
2. Patient who is currently pregnant and enrolled in one of the following SK life science studies: YKP3089C013, YKP3089C017 or YKP3089C021 may enter the EAP program.
3. Written informed consent signed by the patient or legal guardian prior to entering the EAP in accordance with the ICH GCP guidelines. If the written informed consent is provided by the legal guardian because the patient is unable to do so, a written or verbal consent from the patient must also be obtained.

EXCLUSION CRITERIA

1. Patients that have previously discontinued for any reason from studies YKP3089C013, YKP3089C017 and YKP3089C021.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.